CLINICAL TRIAL: NCT00404066
Title: Phase II Neoadjuvant Chemotherapy Trial in Clinical Stage II/III Her2Neu Positive Breast Cancer With Sequential AC -> Docetaxel With Concurrent Dual EGFR Kinase Blockade by GW572016 (Lapatinib) Followed by 1 Year Adjuvant Trastuzumab
Brief Title: Phase 2 Neoadjuvant Doxorubicin and Cyclophosphamide -> Docetaxel With Lapatinib in Stage II/III Her2Neu+ Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: George Albert Fisher (Other)
Collaborators: GlaxoSmithKline (Industry); Sanofi (Industry)
Responsible Party: Sponsor-Investigator, George Albert Fisher, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-03518; BRSADJ0002 (Other: OnCore)
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Doxorubicin; Cyclophosphamide; Docetaxel; pegfilgrastim; Filgrastim; Granulocyte Colony-Stimulating Factor; Dexamethasone; Calcium Dobesilate; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Chemotherapy (Experimental): Doxorubicin (Adriamycin) + cyclophosphamide (Cytoxan) with pegfilgrastim or filgrastim growth factor support every 2 weeks for 4 cycles, followed by docetaxel + lapatinib for four 21-day cycles, followed by surgery. Dexamethasone was administered twice-a-day for 3 days, starting 24 hours before the docetaxel infusions. After surgery +/- radiation, participants may receive trastuzumab (Herceptin) for a year.
  Interventions: Drug: Lapatinib; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Pegfilgrastim; Drug: Filgrastim; Drug: Dexamethasone; Drug: Trastuzumab

INTERVENTIONS:
Drug: Lapatinib — 1250 mg, tablets, oral daily during treatment with docetaxel (3-week cycles x 4 cycles)
  Other Names: GW572016
Drug: Doxorubicin — 60 mg/m2, intravenously every 2 weeks for 4 cycles. Given as first treatment with cyclophosphamide.
  Other Names: Adriamycin; Adriablastin
Drug: Cyclophosphamide — 600 mg/m2, intravenously every 2 weeks for 4 cycles. Given as first treatment with doxorubicin.
  Other Names: Cytoxan; ASTA
Drug: Docetaxel — 100 mg/m2, intravenously every 3 weeks for 4 cycles (after treatment cycles of doxorubicin and cyclophosphamide
  Other Names: Taxotere
Drug: Pegfilgrastim — 6 mg, subcutaneously on day 2 of all cytotoxic chemotherapy treatments.
  Other Names: Neulasta
Drug: Filgrastim — 300 or 480 mcg, subcutaneously on days 3 to 10 after cytotoxic chemotherapies.
  Other Names: Neupogen; Granulocyte Colony-Stimulating Factor (G-CSF)
Drug: Dexamethasone — 8 mg, oral taken twice a day for 3 days starting 24 hours before docetaxel
  Other Names: Adexone
Drug: Trastuzumab — Loading dose 8 mg/kg, then 6 mg/kg, intravenously every 3 weeks for 1 year
  Other Names: Herceptin

SUMMARY:
This trial combines dose dense chemotherapy with doxorubicin and cyclophosphamide (AC) followed by standard, every 3 week docetaxel and GW572016 (lapatinib) for neoadjuvant treatment of Her2neu positive stage II/III breast cancer. The purpose of the study was to determine whether lapatinib combined with chemotherapy was safe and resulted in an increase in pathologic complete response rates.

DETAILED DESCRIPTION:
Lapatinib acts as a dual inhibitor of both epidermal growth factor receptor (EGFR) and ErbB-2 (Her2/neu) tyrosine kinase activity. EGFR and ErbB2 receptors are frequently over-expressed or altered in human cancers including breast cancer. This study plans to determine the antitumor activity of this regimen and its effectiveness preventing tumor growth and spread.

Neoadjuvant chemotherapy which achieves pathologic complete responses (pCR) has been shown to predict improved long-term survival and serves as a surrogate for clinical outcome. By using this primary endpoint we can obtain statistical data with smaller patient numbers and at a lower overall cost. Additionally, we hope to correlate clinical and radiologic outcomes with gene expression data.

ELIGIBILITY:
INCLUSION CRITERIA

* Female
* Histologically-confirmed Her2neu positive breast cancer, by either Immunohistochemistry (IHC) 3+ or Fluorescence In Situ Hybridization (FISH)+
* Stage II/III breast cancer including any large primary tumor (> 2 cm), tumors of any size associated with skin or chest wall involvement, tumors of any size with axillary lymph node involvement, (T2-T4, N0-N2) and those with ipsilateral subclavicular or supraclavicular lymph nodes).
* At least one bi-dimensional, measurable indicator lesion.
* Between 18 and 70 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 / Karnofsky ≥ 60% at screening and on the first day of treatment.
* Informed consent must be obtained prior to registration.
* Cardiac ejection fraction within the institutional range of normal as measured by multigated acquisition (MUGA) or echocardiography (ECHO) scan.
* Absolute neutrophil count > 1,500/mm³
* Hemoglobin > 8.0 g/dL
* Platelet count > 100,000/mm³
* Creatinine within normal institutional limits
* Total Bilirubin equal to or less than institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST); alanine aminotransferase (ALT); and alkaline phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values (AST or ALT) should be used.
* Eligibility of patients receiving medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of GW572016 will be determined following review of their use by the Principal Investigator

  * Antacid use is prohibited 1 hour before and 1 hour after GW572016 dosing.
  * All herbal (alternative) medicines are prohibited.
  * Medications prohibited during the administration of lapatinib .
* Women of child-bearing potential must have negative pregnancy test and must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation.
* Peripheral neuropathy: must be < grade 1
* Able to swallow and retain oral medication

EXCLUSION CRITERIA

* Evidence of disease outside the breast or chest wall, except for ipsilateral axillary , supraclavicular, or infraclavicular lymph nodes.
* Prior chemotherapy, immunotherapy, or hormonal therapy for breast cancer.
* More than 3 months between histologic diagnosis and registration on this study.
* History of other malignancy within the last 5years, except curatively treated basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Psychological, familial, sociological or geographical conditions which do not permit weekly medical follow-up and compliance with the study protocol. Those who are medically-unstable, including but not limited to active infection, acute hepatitis, deep vein thrombosis requiring anticoagulant therapy, gastrointestinal bleeding, uncontrolled hypercalcemia, uncontrolled diabetes, dementia, seizures, superior vena cava syndrome, and those whose circumstances do not permit completion of the study or the required follow-up.
* Congestive heart failure, abnormal left ventricular ejection fraction (LVEF), angina pectoris, uncontrolled cardiac arrhythmias, or other significant heart disease, or who have had a myocardial infarction within the past year.
* Pregnant or lactating
* Of childbearing potential and not employing adequate contraception
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016.
* HIV-positive and receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with lapatinib. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
* GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* History of severe hypersensitivity reaction to taxotere or other drugs formulated with polysorbate 80.
* Current active hepatic or biliary disease (with exception of patients with Gilberts syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment ).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Fisher, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Chemotherapy
Started | 21 (1 subject started but withdrew after adriamycin+cytoxan, but before study drugs lapatinib+docetaxel.)
Completed | 18
Not Completed | 3
Not completed — Withdrawal by Subject - Pre-treatment | 1
Not completed — Withdrawal by Subject - Adverse event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Histology [Count of Participants; unit: Participants]
  Ductal | 21
  Lobular | 0
Tumor Size [Count of Participants; unit: Participants] — Tumors were staged according to T stage:
  * T1: Malignancy is ≤ 20 millimeters (mm) at the widest spot
  * T2: Malignancy is > 20 mm but ≤ 50 mm
  * T3: Malignancy is > 50 mm
  * T4: Metastasized to chest wall and/or skin
  Participants
    T1 (≤ 20 mm at widest) | 0
    T2 (> 20 mm but ≤ 50 mm) | 9
    T3 (> 50 mm) | 9
    T4 (metastatic to chest wall / skin) | 3
Nodal involvement [Count of Participants; unit: Participants] — Tumors were staged by lymph node involvement according to the following criteria.
  * N1: The cancer has spread to 1 to 3 axillary, or underarm, lymph nodes under the arm, and are ≥ 2 mm in size.
  * N2: The cancer has spread to 4 to 9 axillary lymph nodes, OR has spread to internal mammary lymph nodes
  * N3: The cancer has spread to ≥ 10 lymph nodes, OR has spread to both axillary and internal mammary lymph nodes
  Participants
    N1 (few lymph nodes) | 3
    N2 (moderate number of lymph nodes) | 13
    N3 (many lymph nodes) | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathologic Complete Response (pCR)
Description: Pathologic Complete Response (pCR) rate, assessed as no evidence of invasive disease in excised surgical specimens of breast and/or axilla, in participants who received at least 1 cycle of docetaxel and lapatinib and at least one follow-up evaluation.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 18
percentage of participants | 38.9

2. Secondary Outcome: Disease-free Survival (DFS)
Description: Disease-free survival (DFS) is expressed as the percentage of participants who were disease-free and alive at the time of analysis.
Time Frame: 42 months (median follow-up)
Population: DFS is reported as the number and percentage of participants who were alive and disease-free at the time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 18
Participants | 16

ADVERSE EVENTS:
Time Frame: up to 5 years
Arm/Group | Neoadjuvant Chemotherapy
All-Cause Mortality (participants affected / at risk) | 2/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemotherapy (N=21)
Irregular menses (Reproductive system and breast disorders) | 20 (20)
Hand-foot-skin reactions (Skin and subcutaneous tissue disorders) | 20 (20)
Nausea (Gastrointestinal disorders) | 14 (14)
Nail bed changes (General disorders) | 14 (14)
Dysphagia (mouth pain) (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Adrenal insufficiency (Metabolism and nutrition disorders) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Anemia (Blood and lymphatic system disorders) | 17 (17)
Mucositis (Gastrointestinal disorders) | 2 (2)
Arthralgia (joint pain) (General disorders) | 1 (1)
Pain, general (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No